CLINICAL TRIAL: NCT02088840
Title: A Prospective, Multicenter Survey of Severe Infections by Gram Negative Bacteria in Patients Submitted to Autologous and Allogeneic Stem Cell Transplant.
Brief Title: Survey of Severe Infections by Gram Negative Bacteria in Patients Submitted to Stem Cell Transplant
Acronym: GITMO-SIGNB
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Other Study IDs: SIGNB-GITMO-AMCLI-Survey
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Complications of Organ Transplant Stem Cells; Gram-Negative Bacterial Infections
Keywords: SIGNB; severe infections gram negative bacteria; stem cell transplant
MeSH Terms: conditions — Gram-Negative Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stem cell tranplant: All patients undergoing autologous or allogeneic stem cell tranplant for any underlying disease

SUMMARY:
All patients undergoing autologous or allogeneic stem cell transplant (SCT) for any underlying disease will be monitored for severe infections by gram negative bacteria (SIGNB) during the engraftment period. The follow up will be stopped at 4 months from the day of transplant. About 50 transplant centers will be involved in the study.

DETAILED DESCRIPTION:
Severe Infections by Gram Negative Bacteria (SIGNB) remain an important cause of morbidity and mortality in patients submitted to stem cell transplant particularly during engraftment while patients suffer of profound and prolonged neutropenia or during subsequent neutropenia periods related to loss of engraftment or viral infections. Epidemiology of severe infections by gram negative bacteria in stem cell transplant patients has varied in the last decades due to the increasing use of highly immunosuppressive stem cell transplant procedures, and in relation to global epidemiological phenomena involving several populations of immunocompromised patients including those submitted to stem cell transplant.

The epidemiological evolution of severe infections by gram negative bacteria in immunocompromised patients is represented also by the emergence of infections caused by Gram-negative bacilli, in particular enterobacteria, resistant to several antimicrobials. Such pattern of susceptibility to antibacterial agents represents a challenging issue in the currents strategies of the use of antibiotics in prophylaxis or therapy.

Despite an increasing attention to the clinical and therapeutic aspects of infection in stem cell transplant recipients, contrasting data are available on the incidence, microbiologic characteristics and clinical outcome of Severe Infections by Gram Negative Bacteria in this population.

Management of patients submitted to stem cell transplant is frequently complicated by Severe Infections by Gram Negative Bacteria which may represent an obstacle to the transplant procedure. Severe Infections by Gram Negative Bacteria caused by microorganisms resistant to betalactamic antibiotics, which are the golden standard in the empirical antibacterial therapy of febrile neutropenia, represent a challenging problem. A revision of the antibacterial strategies and the consideration of new molecules with different antibacterial mechanism of action should be considered in the light of the emerging epidemiology. Antimicrobial prophylaxis, diagnostic approaches and antimicrobial therapy should be adapted to the infectious risk of the transplant population according to stem cell source, conditioning regimen and also to the infectious history before transplant. A crucial problem in the definition of these strategies is represented by the continuous change in the epidemiological patterns of infections as a result of the modification of risk factors in the transplant population and of the global epidemiology of hospital and community acquired infections. In particular the emergence of antibiotic resistant enterobacteria represents a serious problem which dramatically impacts on the antibacterial prophylaxis and treatments choices.

The Investigator think that a continuous epidemiology survey is required in order to better define proper prevention, diagnostic and treatment approaches. A common problem in the infections control in immunocompromised populations is represented by the lack of epidemiological consciousness in the single centres and its relationship with the local policy in the use of antibacterial drugs. A prospective, multicenter survey of Severe Infections by Gram Negative Bacteria by antibiotic resistant pathogens, in particular enterobacteria, may be a useful tool to evaluate the epidemiological patterns of infections, their impact on the overall survival, and a critical analysis of the use of antibacterial drugs.

The Investigator of this study think that the results of this survey may offer precious indications for the timely update of the prophylaxis, diagnosis and treatment strategies of Severe Infections by Gram Negative Bacteria in patients undergoing a stem cell transplant procedure.

An important aspect of this study is represented by the involvement of both stem cell transplant and microbiology Italian societies, the GITMO Gruppo Italiano per il Trapianto di Midollo Osseo, cellule staminali emopoietiche e terapia cellulare and the AMCLI Associazione Microbiologi Clinici Italiani respectively, as a "joint venture" in the study of the clinical and microbiological aspects of Severe Infections by Gram Negative Bacteria in the autologous and allogeneic stem cell transplant populations. Investigators of both GITMO and AMCLI are involved in the design, writing and monitoring of the study and for each participating transplant center a clinician, responsible for the clinical data, and a microbiologist, responsible for the microbiological data, will be provided.

The general objectives of this study are to prospectively evaluate the epidemiology of Severe Infections by Gram Negative Bacteria by antibiotic resistant pathogens in autologous and allogeneic stem cell transplant patients during the engraftment period.

All consecutive patients submitted to autologous or allogeneic stem cell transplant for any underlying disease in about 50 Italian transplant centers will be prospectively monitored for severe infections by gram negative bacteria during the engraftment period. The follow up will be stopped at 4 months from the day of transplant. Risk factors, incidence and prognostic factors of Severe Infections by Gram Negative Bacteria will be evaluated in the overall population and in subpopulations according to different transplant characteristics. Data on in vitro susceptibility patterns of the microorganisms and on the antibacterials used in prophylaxis and therapy will be collected.

Descriptive analyses will be performed for all Severe Infections by Gram Negative Bacteria cases occurring among patients enrolled in this study.

The study will be conducted in accordance with the ethical principles derived from the Declaration of Helsinki, the CGP and regulations.

In this study the investigators will use the E-CRF in apposite web site. Data will be collected in E-CRF (electronic case report form) for the registration of clinical data through a special web portal dedicated to the study.

Investigators are responsible for the preparation and storage of clinical data concerning the clinical trial in accordance with ICH guidelines for good clinical practice. Access to clinical data should be reserved exclusively to authorized personnel. Investigators will have to verify and ensure the strict confidentiality of records that could identify patients in compliance with standards on privacy and personal data in accordance with Italian legislation. On data collection forms (and related documentation) patients should be uniquely identified by date of birth and the code of enrolment. The full name of the patient will never be used in any communication and / or correspondence. Will be required direct access to the patient's original medical records for verification and monitoring of clinical data. The investigators are obliged to inform patients that their medical records could be verified, without breach of confidentiality of personal data. Investigators will have to allow monitoring of clinical data related to the study, the revisions IRB / IEC and inspections by regulatory authorities in accordance with Italian legislation, providing direct access to the medical records of patients.

The national coordination of the study is carried out by the Office of Clinical Trials GITMO. The Office of Clinical Trials GITMO will act as the Data Management Center and quality control, providing for data management and administrative support throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients submitted to autologous or allogeneic SCT at the Centers participating to the survey Signed written informed consent according to IGH/EU/GCP and national local laws.

Without age limit

Exclusion Criteria:

Patients who did not sign written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing autologous or allogeneic Stem Cell Transplant for any underlying disease will be monitored for SIGNB during the engraftment period.
Sampling Method: Non-Probability Sample
Enrollment: 2769 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
incidence of each type of Severe Infections by Gram Negative Bacteria | 4 months by stem cell transplant
  To estimate the incidence of each type of Severe Infections by Gram Negative Bacteria , in particular by antibiotic resistant isolates, documented during the engraftment period in patients submitted to autologous and allogeneic stem cell transplant.

SECONDARY OUTCOMES:
incidence particularly of Severe Infections by Gram Negative Bacteria | 4 months by stem cell transplant
  To assess the incidence of Severe Infections by Gram Negative Bacteria particularly those caused by antibiotic resistant enterobacteria in subgroups of patients undergoing autologous or allogeneic stem cell transplant.
risk factors | 4 month by stem cell transplant
  To assess the risk factors of Severe Infections by Gram Negative Bacteria particularly those caused by antibiotic resistant enterobacteria in autologous and allogeneic Stem cell CT transplant
prognostic factors | 4 month by stem cell transplant
  To assess the prognostic factors of Severe Infections by Gram Negative Bacteria particularly those caused by antibiotic resistant enterobacteria in autologous and allogeneic Stem cell CT transplant
overall mortality for SIGNB | 3 months from the Severe Infections by Gram Negative Bacteria
  To assess the overall Severe Infections by Gram Negative Bacteria and attributable mortality at 3 months from the SIGNB
overall survival for SIGNB from transplant | 4 months from transplant
  To assess the impact of SIGNB on the overall survival at 4 months from transplant in autologous and allogeneic Stem Cell Transplantation
susceptibility pattern to antimicrobials of microorganisms | 4 month by stem cell transplant
  To evaluate the susceptibility pattern to antimicrobials of microorganisms causing Severe Infections by Gram Negative Bacteria with particular attention to enterobacteria with particular attention to the resistance phenotypes
antibacterial strategies | 4 month by stem cell transplant
  To describe the antibacterial strategies (in prophylaxis and therapy) employed in the various centers and in the various categories of patients particularly for the management of antibiotic resistant enterobacteria
local strategy | 4 month by stem cell transplant
  To evaluate the impact of a local strategy in the use of antibiotics on the epidemiology of Severe Infections by Gram Negative Bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Girmenia, MD, Principal Investigator — Policlinico Umberto I - Rome
Locations (54):
- Italy (54):
  - FPO Irccs, Candiolo, Torino
  - Azienda Ospedaliera SS Antonio e Biagio, Alessandria
  - Clinica di Ematologia - Università Politecnica delle Marche, Ancona
  - Ospedale Mazzoni, Ascoli Piceno
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Divisione di Ematologia - Ospedali Papa Giovanni XXIII, Bergamo
  - Ospedale San Orsola, Bologna
  - AO Spedali Civili di Brescia- USD - TMO Adulti, Brescia
  - Spedali Civili, Brescia
  - Ospedale Binaghi, Cagliari
  - Ospedale Ferrarotto - Ematologia, Catania
  - Ospedale Civile USL 8, Civitanova Marche
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Cattedra di Ematologia - Azienda Ospedaliera di Careggi, Florence
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, Foggia
  - AOU IRCCS San Martino - IST, Genova
  - Ospedale Gaslini, Genova
  - Divisione di Ematologia - Istituto Nazionale dei Tumori, Milan
  - IEO, Milan
  - Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - A.O.U. Policlinico Federico II, Napoli
  - INT IRCCS Fondazione Pascale, Napoli
  - Ospedale Maggiore della Carità, Novara
  - AO Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Dipartimento Oncologico La Maddalena, Palermo
  - CTMO Università, Parma
  - Fondazione IRCCS San Matteo, Pavia
  - Dipartimento di Ematologia - IRCCS Policlinico S. Matteo - Università di Pavia, Pavia
  - Dip. Medicina Clinica e Sperimentale, Perugia
  - Dip. di Ematologia - Unità di Terapia Intensiva Ematologica per il Trapianto Emopoietico - Ospedale Civile di Pescara, Pescara
  - Ospedale G. Da Saliceto di Piacenza, Piacenza
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - Ospedale Infermi, Rimini
  - Irccs Crob, Rionero in Vulture
  - A.O. San Camillo, Roma
  - Campus biomedico, Roma
  - Cattedra di Ematologia - Policlinico, Roma
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - Istituto Regina Elena IFO, Roma
  - Ospedale Bambin Gesù, Roma
  - Ospedale San Giovanni, Roma
  - Ospedale Sant'Andrea, Roma
  - Ospedale Santo Eugenio, Roma
  - Policlinico Universitario Tor Vergata, Roma
  - Dipartimento di Oncologia Medica ed Ematologia - Istituto Clinico Humanitas, Rozzano (MI)
  - Ospedale Moscati, Taranto
  - Azienda ospedaliera Città della Salute e della Scienza, Torino
  - Centro Trapianti Metropolitano, Torino
  - Ospedale Gonzaga, Torino
  - UOC Ematologia, Treviso
  - A.O. Santa Maria della Misericordia, Udine
  - Policlinico GB Rossi, Verona
  - Ospedale S. Bortolo-Divisione Ematologia, Vicenza

REFERENCES:
- [Derived] Girmenia C, Bertaina A, Piciocchi A, Perruccio K, Algarotti A, Busca A, Cattaneo C, Raiola AM, Guidi S, Iori AP, Candoni A, Irrera G, Milone G, Marcacci G, Scime R, Musso M, Cudillo L, Sica S, Castagna L, Corradini P, Marchesi F, Pastore D, Alessandrino EP, Annaloro C, Ciceri F, Santarone S, Nassi L, Farina C, Viscoli C, Rossolini GM, Bonifazi F, Rambaldi A; Gruppo Italiano Trapianto di Midollo Osseo (GITMO) and Associazione Microbiologi Clinici Italiani (AMCLI). Incidence, Risk Factors and Outcome of Pre-engraftment Gram-Negative Bacteremia After Allogeneic and Autologous Hematopoietic Stem Cell Transplantation: An Italian Prospective Multicenter Survey. Clin Infect Dis. 2017 Nov 13;65(11):1884-1896. doi: 10.1093/cid/cix690. PMID 29020286